CLINICAL TRIAL: NCT06762496
Title: Development and Testing of a Patient's Decision Aid for Early Breast Cancer: a New Tool to Promote Patient's Engagement in Their Healthcare Process
Brief Title: A New Tool to Promote Patient's Engagement in Their Healthcare Process
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4841
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-11

CONDITIONS: Breast Carcinoma; Breast Cancer Stage I; Breast Cancer Stage II
Keywords: early breast cancer; Patient Decision; engagement
MeSH Terms: conditions — Breast Neoplasms | interventions — Health Personnel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stakeholders: physicians involved in the diagnosis and treatment decision for patients with early breast cancer (10 oncologists, 10 breast surgeons, and 10 breast radiologists specifically).
  Interventions: Other: Healthcare professionals
- Patients PDA group: Participants randomized in this group will receive via mail the final version of the PDA and a Qualtrics link with a battery of questionnaires
  Interventions: Other: Patients PDA group
- Patients control group: Patients randomized in this group will receive only the online link with the battery of questionnaires.
  Interventions: Other: Patients control group

INTERVENTIONS:
Other: Healthcare professionals — healthcare professionals (HCPs) targeted, including team members: we will involve 30 physicians (who are involved in the process of care towards patients with early breast cancer (10 oncologists, 10 breast surgeon, and 10 breast radiologists specifically) for the semi-structured interviews
  Groups: Stakeholders
Other: Patients PDA group — Participants will receive via mail the final version of the PDA and a Qualtrics link with a battery of questionnaires
  Groups: Patients PDA group
Other: Patients control group — Participants will receive only the online link with the battery of questionnaires
  Groups: Patients control group

SUMMARY:
Women diagnosed with early-stage breast cancer need to make a decision about the therapeutic treatment to undertake. Since multiple factors can influence this decision, it is necessary to develop a decision-making support tool to assist them in making this choice.

Main Objective: To develop a decision-making support tool for determining the treatment to undertake for women diagnosed with early-stage breast cancer and test its effectiveness on an experimental group.

DETAILED DESCRIPTION:
Women with any type of early breast cancer (0-2A stages) will be recruited at Istituto Europeo di Oncologia (IEO). 170 patients with early breast cancer and 30 clinicians involved in the present project will directly benefit from better-provided care, an increase in patients' knowledge and management of their oncological symptoms, an improved patient-and-doctor relationship, and a reduction of hospital economic costs.

Our interdisciplinary team will include breast cancer patients, oncologists, surgeons, psychologists, radiologists, , and nurses. All members of our team will play an active role in the most important phases of our data-driven project development cycle. A patient-centered approach will allow us to ensure their active participation from the design phase to the dissemination phase of the project.

This present research project will be based on two different prospective studies: a first study based on patients already treated for breast cancer and a second study with patients newly diagnosed with early breast cancer.

Semi structured interviews will be used in the first study, while newly diagnosed women in the second study will be asked to fill in an online battery of questionnaires in three different times (T0: one week after the first consultation; T1: a month later the first medical consultation; T2: three months later the first medical consultation) to assess the possible impact of using the Patient Decision Aids (PDA) on the doctor-patient communication and shared decision-making (SDM) process.

This project will follow a multi-step approach and will be therefore divided into different developmental phases, within which specific objectives will need to be reached in order to move forward.

Assessment measures throughout the protocol include: AttrakDiff; SUS, a 38-item specific questionnaire that measures satsifaction with PDA, PHQ-9, STAI, SDMQ9, Distress thermometer, EORTC-QLQ.C30, EORT-QLQ-BR23. Any further material used for qualitative assessment will be be made available upon reasonable request.

ELIGIBILITY:
Inclusion Criteria:

* be 18 or older;
* have received/receive diagnosis of resectable breast cancer in the early stage;
* women treated or who will undergo oncological treatment for early breast cancer;
* demonstrate the absence of psychopathological features.
* be willing and able to provide written informed consent/assent for the trial

Exclusion Criteria:

* breast cancer patients who showed physical or psychological issues, as well as cognitive impairments that prohibited their participation in this type of study;
* neurological or psychiatric disorders that may compromise the patients' ability to take part in the study.
* Distant metastases from breast cancer or locally advanced/unresectable disease
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Number of healthcare professionals (HCPs) targeted, including team members: we will involve 30 physicians (who are involved in the process of care towards patients with early breast cancer (10 oncologists, 10 breast surgeon, and 10 breast radiologists specifically) for the semi-structured interviews. Moreover, about 10-12 professionals will take part in the steering committee.
  Number of Patients affected: we will involve patients with early breast cancer for a total of 170 participants, considering all phases of the present project.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Development of an ad hoc Patient Decision Aid (PDA) | 3 months
  Patients in the Intervention group will receive via mail the final version of the PDA and a battery of questionnaires.
  Patients in the Control group will receive only the online link with the battery of questionnaires.
  In both the experimental and the control group, questionnaires will be administered one week after the first medical consultation (T0), one month later the first medical consultation (T1), and three months later the first medical consultations (T2).
  The difference between T1 and T0 and T2 and T0 will be calculated for each endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Dissemination of results will follow typical academic pathways, such as conference abstracts and peer-reviewed journals
Supporting Information: Study Protocol
Time Frame: Jan 2025 - Sep 2026